CLINICAL TRIAL: NCT02315547
Title: Guangzhou Institute of Respiratory Disease
Brief Title: Sputum Microbiota and the Association With Clinical Parameters in Steady-state, Acute Exacerbation and Convalescence of Bronchiectasis
Acronym: BISER-2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Principal Investigator, Weijie Guan, physician, Guangzhou Institute of Respiratory Disease
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GIRD-20141208-GWJ
Record Dates: First submitted 2014-12-08; First posted 2014-12-12 (Estimated); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Bronchiectasis
Keywords: Microbiota; Airway infection; Bronchiectasis; Airway inflammation; Oxidative stress; Matrix metalloproteinase
MeSH Terms: conditions — Bronchiectasis | interventions — Anti-Bacterial Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Antibiotics (Other): Patients will be given antibiotics based on sputum microbiology during steady-state bronchiectasis. The methodology has been described in the British Thoracic Society guideline [16]. Briefly, for first-line therapy, patients isolated with Hemophilus influenzae, Hemophilus parainfluenzae, Streptoccus pneumoniae and Moraxella catarrhalis at baseline will be treated with amoxicillin clavulanate potassium (625mg bid); patients isolated with Klebsela pneumonae or Pseudomonas aeruginosa at baseline will be treated with fluoroquinolones. Levofloxacin (500mg qd) will be empirically employed for antibiotic treatment in those who tested negative to sputum microbiology. Severe BEs could be prescribed with intravenous antibiotics therapy at the discretion of study investigators, either in the out-patient department or hospitalized for intensive systemic treatment. Hospitalized patients will not be included in the exacerbation cohort.
  Interventions: Drug: Antibiotics

INTERVENTIONS:
Drug: Antibiotics — Patients will be given antibiotics based on sputum microbiology during steady-state bronchiectasis. The methodology has been described in the British Thoracic Society guideline [16]. Briefly, for first-line therapy, patients isolated with Hemophilus influenzae, Hemophilus parainfluenzae, Streptoccus pneumoniae and Moraxella catarrhalis at baseline will be treated with amoxicillin clavulanate potassium (625mg bid); patients isolated with Klebsela pneumonae or Pseudomonas aeruginosa at baseline will be treated with fluoroquinolones. Levofloxacin (500mg qd) will be empirically employed for antibiotic treatment in those who tested negative to sputum microbiology. Severe BEs could be prescribed with intravenous antibiotics therapy at the discretion of study investigators, either in the out-patient department or hospitalized for intensive systemic treatment. Hospitalized patients will not be included in the exacerbation cohort.

SUMMARY:
Study 1 is a cross-sectional investigation. Patients with clinically stable bronchiectasis (symptoms, including cough frequency, sputum volume and purulence, within normal daily variations) will undergo baseline assessment consisting of history taking, routine sputum culture, 16srRNA pyrosequencing, measurement of sputum inflammatory markers, oxidative stress biomarkers and MMPs, and spirometry. Microbiota taxa will be compared between bronchiectasis patients and healthy subjects.

In study 2, patients inform investigators upon symptom deterioration. Following diagnosis of BEs, patients will undergo the aforementioned assessments as soon as possible. This entails antibiotic treatment, with slightly modified protocol, based on British Thoracic Society guidelines [16]. At 1 week after completion of 14-day antibiotic therapy, patients will undergo convalescence visit.

Study 3 is a prospective 1-year follow-up scheme in which patients participated in telephone or hospital visits every 3 months. For individual visit, spirometry and sputum culture will be performed, and BEs will be meticulously captured from clinical charts and history inquiry, with the final decisions adjudicated following group discussion.

DETAILED DESCRIPTION:
Bronchiectasis is a chronic airway disease characterized by airway infection, inflammation and destruction [1]. Bacteria are frequently responsible for the vicious cycle seen in bronchiectasis. Clinically, potentially pathogenic microorganisms (PPMs) primarily consisted of Hemophilus influenzae, Hemophilus parainfluenzae, Pseudomonas aeruginosa (P. aeruginosa), Staphylococcus aureus, Klebsiella pneumoniae, Streptococcus pneumoniae and Moraxella catarrhalis [1]. These PPMs elicit airway inflammation [2-5] and biofilm formation [6] leading to and oxidative stress [7,8]. However, different PPMs harbor varying effects on bronchiectasis. For instance, P. aeruginosa has been linked to more pronounced airway inflammation and poorer lung function [9,10].

However, it should be recognized that routine sputum bacterial culture techniques could only effectively identify a small proportion of PPMs. The assay sensitivity and specificity could be significantly affected by the duration from sampling to culture, the culture media and environment. Pyrosequencing of the bacterial 16srRNA might offer more comprehensive assessment of the airway microbiota. Based on this technique, Goleva and associates [11] identified an abundance of gram-negative microbiota (predominantly the phylum proteobacteria) which might be responsible for corticosteroid insensitivity. The microbiome of airways in patients with asthma [11,12], idiopathic pulmonary fibrosis [13] and bronchiectasis [14,15] has also been characterized. Furthermore, the association between the "core microbiota" and clinical parameters (i.e., FEV1) has been demonstrated. However, previous studies suffered from relatively small sample size and lack of comprehensive sets of clinical parameters for further analyses.

Bronchiectasis exacerbations (BEs) are characterized by significantly worsened symptoms and (or) signs that warrant antibiotics therapy. The precise mechanisms responsible for triggering BEs have not been fully elucidated, but could be related to virus infection and increased bacterial virulence. However, it should be recognized that antibiotics, despite extensive bacterial resistance, remain effective for most BEs. This at least partially suggested that bacterial infection might have played a major role in the pathogenesis of BEs. Therefore, the assessment of sputum microbiota during steady-state, BEs and convalescence may unravel more insights into the dynamic variation in microbiota compositions and the principal microbiota phylum or species that account for BEs.

In the this study, the investigators seek to perform 16srRNA pyrosequencing to determine: 1) the differences in microbiota compositions between bronchiectasis patients and healthy subjects; 2) association between sputum microbiota compositions and clinical parameters, including systemic/airway inflammation, spirometry, disease severity, airway oxidative stress biomarkers and matrix metalloproteinase; 3) the microbiota compositions in patients who yielded "normal flora (commensals)", in particular those who produced massive sputum daily (>50ml/d); 4) dynamic changes in microbiota compositions during BEs and convalescence as compared with baseline levels; 5) the utility of predominant microbiota taxa in predicting lung function decline and future risks of BEs during 1-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patients of either sex and age between 18 and 85 years

Exclusion Criteria:

1. Patient judged to have poor compliance
2. Female patient who is lactating or pregnant
3. Patients having concomitant severe systemic illnesses (i.e. coronary heart disease, cerebral stroke, uncontrolled hypertension, active gastric ulcer, malignant tumor, hepatic dysfunction, renal dysfunction)
4. Miscellaneous conditions that would potentially influence efficacy assessment, as judged by the investigators
5. Participation in another clinical trial within the preceding 3 months

Inclusion criteria for healthy subjects include all of the above criteria except for known respiratory diseases

It is estimated that 120 patients will be recruited in the study. Some of the patients in the BISER study (currently still ongoing, No.: NCT01761214) who are eligible for the current study will undergo assessments de novo, with the index date deemed as the the date of recruitment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-01; Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
relative abundance, diversity and richness of microbiota taxa | Jan 2015 to Dec 2017, up to 3 years
  Sputum microbiota taxa compositions (at phylum and species levels, respectively), including the relative abundance, diversity and richness

SECONDARY OUTCOMES:
Serum inflammatory indices | Jan 2015 to Dec 2017, up to 3 years
  IL-8, TNF-α, WBC and CRP
Sputum sol phase inflammatory biomarkers | Jan 2015 to Dec 2017, up to 3 years
  IL-8 and TNF-α
Sputum sol phase oxidative stress biomarkers or parameters | Jan 2015 to Dec 2017, up to 3 years
  CAT, hydrogen peroxide, superoxide dismutase, MDA
Sputum sol phase matrix metalloproteinases | Jan 2015 to Dec 2017, up to 3 years
  MMP-8, MMP-9, TIMP-1, MMP-9/TIMP-1 ratio
24-hour sputum volume | Jan 2015 to Dec 2017, up to 3 years
  24-hour sputum volume, measured to the nearest 5 ml
Spirometry | Jan 2015 to Dec 2017, up to 3 years
  FEV1, FVC, FEV1/FVC, MMEF
Bronchiectasis Severity Index | Jan 2015 to Dec 2017, up to 3 years
Sputum culture findings | Jan 2015 to Dec 2017, up to 3 years
  normally reported as growth of a predominant potentially pathogenic microorganism or no bacterial growth
Sputum purulence | Jan 2015 to Dec 2017, up to 3 years
  scale 1 to 8
SGRQ total score and the scores of individual domains | Jan 2015 to Dec 2017, up to 3 years
  SGRQ total score and the scores of individual domains

CONTACTS AND LOCATIONS:
Overall Officials: Nan-shan Zhong, MD, Study Chair — State Key Laboraotry of Respiratory Disease
Locations (1):
- Guangzhou Institute of Respiratory Disease, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Pasteur MC, Helliwell SM, Houghton SJ, Webb SC, Foweraker JE, Coulden RA, Flower CD, Bilton D, Keogan MT. An investigation into causative factors in patients with bronchiectasis. Am J Respir Crit Care Med. 2000 Oct;162(4 Pt 1):1277-84. doi: 10.1164/ajrccm.162.4.9906120. PMID 11029331
- [Background] Davies G, Wells AU, Doffman S, Watanabe S, Wilson R. The effect of Pseudomonas aeruginosa on pulmonary function in patients with bronchiectasis. Eur Respir J. 2006 Nov;28(5):974-9. doi: 10.1183/09031936.06.00074605. Epub 2006 Aug 9. PMID 16899482
- [Background] Chmiel JF, Davis PB. State of the art: why do the lungs of patients with cystic fibrosis become infected and why can't they clear the infection? Respir Res. 2003;4(1):8. doi: 10.1186/1465-9921-4-8. Epub 2003 Aug 27. PMID 14511398
- [Background] King PT, Hutchinson PE, Johnson PD, Holmes PW, Freezer NJ, Holdsworth SR. Adaptive immunity to nontypeable Haemophilus influenzae. Am J Respir Crit Care Med. 2003 Feb 15;167(4):587-92. doi: 10.1164/rccm.200207-728OC. Epub 2002 Nov 14. PMID 12433671
- [Background] Sadikot RT, Blackwell TS, Christman JW, Prince AS. Pathogen-host interactions in Pseudomonas aeruginosa pneumonia. Am J Respir Crit Care Med. 2005 Jun 1;171(11):1209-23. doi: 10.1164/rccm.200408-1044SO. Epub 2005 Feb 1. PMID 15695491
- [Background] Starner TD, Zhang N, Kim G, Apicella MA, McCray PB Jr. Haemophilus influenzae forms biofilms on airway epithelia: implications in cystic fibrosis. Am J Respir Crit Care Med. 2006 Jul 15;174(2):213-20. doi: 10.1164/rccm.200509-1459OC. Epub 2006 May 4. PMID 16675778
- [Background] Horvath I, Loukides S, Wodehouse T, Kharitonov SA, Cole PJ, Barnes PJ. Increased levels of exhaled carbon monoxide in bronchiectasis: a new marker of oxidative stress. Thorax. 1998 Oct;53(10):867-70. doi: 10.1136/thx.53.10.867. PMID 10193374
- [Background] Angrill J, Agusti C, De Celis R, Filella X, Rano A, Elena M, De La Bellacasa JP, Xaubet A, Torres A. Bronchial inflammation and colonization in patients with clinically stable bronchiectasis. Am J Respir Crit Care Med. 2001 Nov 1;164(9):1628-32. doi: 10.1164/ajrccm.164.9.2105083. PMID 11719301
- [Background] Ryall B, Davies JC, Wilson R, Shoemark A, Williams HD. Pseudomonas aeruginosa, cyanide accumulation and lung function in CF and non-CF bronchiectasis patients. Eur Respir J. 2008 Sep;32(3):740-7. doi: 10.1183/09031936.00159607. Epub 2008 May 14. PMID 18480102
- [Background] Evans SA, Turner SM, Bosch BJ, Hardy CC, Woodhead MA. Lung function in bronchiectasis: the influence of Pseudomonas aeruginosa. Eur Respir J. 1996 Aug;9(8):1601-4. doi: 10.1183/09031936.96.09081601. PMID 8866579
- [Background] Goleva E, Jackson LP, Harris JK, Robertson CE, Sutherland ER, Hall CF, Good JT Jr, Gelfand EW, Martin RJ, Leung DY. The effects of airway microbiome on corticosteroid responsiveness in asthma. Am J Respir Crit Care Med. 2013 Nov 15;188(10):1193-201. doi: 10.1164/rccm.201304-0775OC. PMID 24024497
- [Background] Marri PR, Stern DA, Wright AL, Billheimer D, Martinez FD. Asthma-associated differences in microbial composition of induced sputum. J Allergy Clin Immunol. 2013 Feb;131(2):346-52.e1-3. doi: 10.1016/j.jaci.2012.11.013. Epub 2012 Dec 23. PMID 23265859
- [Background] Garzoni C, Brugger SD, Qi W, Wasmer S, Cusini A, Dumont P, Gorgievski-Hrisoho M, Muhlemann K, von Garnier C, Hilty M. Microbial communities in the respiratory tract of patients with interstitial lung disease. Thorax. 2013 Dec;68(12):1150-6. doi: 10.1136/thoraxjnl-2012-202917. Epub 2013 Aug 14. PMID 23945167
- [Background] Rogers GB, van der Gast CJ, Cuthbertson L, Thomson SK, Bruce KD, Martin ML, Serisier DJ. Clinical measures of disease in adult non-CF bronchiectasis correlate with airway microbiota composition. Thorax. 2013 Aug;68(8):731-7. doi: 10.1136/thoraxjnl-2012-203105. Epub 2013 Apr 6. PMID 23564400
- [Background] Tunney MM, Einarsson GG, Wei L, Drain M, Klem ER, Cardwell C, Ennis M, Boucher RC, Wolfgang MC, Elborn JS. Lung microbiota and bacterial abundance in patients with bronchiectasis when clinically stable and during exacerbation. Am J Respir Crit Care Med. 2013 May 15;187(10):1118-26. doi: 10.1164/rccm.201210-1937OC. PMID 23348972
- [Background] Pasteur MC, Bilton D, Hill AT; British Thoracic Society Bronchiectasis non-CF Guideline Group. British Thoracic Society guideline for non-CF bronchiectasis. Thorax. 2010 Jul;65 Suppl 1:i1-58. doi: 10.1136/thx.2010.136119. PMID 20627931
- [Background] Chalmers JD, Goeminne P, Aliberti S, McDonnell MJ, Lonni S, Davidson J, Poppelwell L, Salih W, Pesci A, Dupont LJ, Fardon TC, De Soyza A, Hill AT. The bronchiectasis severity index. An international derivation and validation study. Am J Respir Crit Care Med. 2014 Mar 1;189(5):576-85. doi: 10.1164/rccm.201309-1575OC. PMID 24328736
- [Background] Laszlo G. Standardisation of lung function testing: helpful guidance from the ATS/ERS Task Force. Thorax. 2006 Sep;61(9):744-6. doi: 10.1136/thx.2006.061648. PMID 16936234
- [Background] Zheng J, Zhong N. Normative values of pulmonary function testing in Chinese adults. Chin Med J (Engl). 2002 Jan;115(1):50-4. PMID 11930658
- [Background] Fodor AA, Klem ER, Gilpin DF, Elborn JS, Boucher RC, Tunney MM, Wolfgang MC. The adult cystic fibrosis airway microbiota is stable over time and infection type, and highly resilient to antibiotic treatment of exacerbations. PLoS One. 2012;7(9):e45001. doi: 10.1371/journal.pone.0045001. Epub 2012 Sep 26. PMID 23049765